CLINICAL TRIAL: NCT04222751
Title: Static Muscular Stretching for Treatment of Peripheral Artery Disease
Brief Title: Static Muscular Stretching for Treatment of PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emily Pritchard, PI, Florida State University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-005234 Mayo; NCT04197609 (obsolete NCT alias)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stretch Group (Experimental): Subjects assigned to this group will be instructed on how to wear the device to produce the appropriate amount of dorsiflexion (stretch). Splint devices will be worn at the assigned angle 5 days/week, 30 minutes/day, for 4 weeks. ABI, muscle oxygenation, and walking distance will be assessed pre/post stretching. Other health surveys will be administered.
  Interventions: Device: Ankle Splint
- No Stretch Group (Placebo Comparator): Subjects assigned to this group will wear the splints but instructed to wear the device in a position that produces no stretch. Splint devices will be worn at the assigned angle 5 days/week, 30 minutes/day, for 4 weeks. ABI, muscle oxygenation, and walking distance will be assessed pre/post stretching. Other health surveys will be administered.
  Interventions: Device: Ankle Splint

INTERVENTIONS:
Device: Ankle Splint — Ankle splint will be slightly modified from the commercial form to include a pneumatic air cell secured under the forefoot below the splint's padded lining. This replaces the foam wedge provided by the manufacturer, allowing a gradual adjustment of the forefoot/toe region.

SUMMARY:
Patients with peripheral arterial disease (PAD) often have walking impairment due to insufficient oxygen supply to skeletal muscle. The investigator's pilot study in PAD patients has shown that endothelial function and walking distance improve with regular static muscle stretching. Therefore, the purpose of this study is to determine whether prescriptive muscle stretching improves muscle oxygenation and walking ability in PAD patients. This is a single-blinded study in 40 patients with stable symptomatic PAD. Patients assigned to the stretch group will use ankle splints (both legs) to perform static muscle stretching for 4 weeks (ankle dorsiflexion applied 30 min/d, 5 days/wk). Patients assigned to the control group will also wear the ankle splints daily but without invoking any dorsiflexion, i.e., without stretching. Measurements will consist of ankle-brachial index (ABI) at rest and post-exercise, skeletal muscle oxygenation (evaluated with near-infrared spectroscopy (NIRS)), and 6 minute walk test (6MWT), performed at baseline and after 4 weeks of stretching (or control splint placement). In addition, NIRS will be used to evaluate muscle oxygenation while patients are wearing the splint device in order to quantitatively prescribe the angle of dorsiflexion that provides optimum stretch and deoxygenation of the calf muscles without causing pain. Primary outcomes include increased muscle oxygenation during exercise and walking distance after 4 weeks of static muscle stretching. Results from this study will be used to support funding applications for a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 40+
* A resting ankle-brachial index (ABI) of 0.90 or less in either leg
* Stable disease (PAD) for a minimum of 3-months

Exclusion Criteria:

* Habitual exercise (30 minutes of continuous activity for 3 or more days per week)
* Cardiovascular rehabilitation program during the past 3 months
* Below or above-knee amputation, critical limb ischemia (ulceration or gangrene)
* Leg pain at rest
* Cardiorespiratory disease
* Diabetes
* Major surgery or lower extremity revascularization during the previous 3 months
* Major medical illness treatment during the prior 12 months
* Central neurological disease
* Limited ankle or knee joint range of motion
* Requirement of oxygen with activity or exercise
* More than a class II New York Heart Association level of heart failure
* Wheelchair confinement, or inability to walk
* Cognitive disorder
* Vasculitis problem including Takayasu's arteritis, Buerger's disease, collagen disease or Raynaud's disease

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Oxygenation | 4 weeks
  Noninvasive assessment via NIRS monitor
Change in Continuous Walking Distance | 4 weeks
  Assessed by 6-minute walking test
Change in Total Walking Distance | 4 weeks
  Assessed by 6-minute walking test

CONTACTS AND LOCATIONS:
Overall Officials: Judy Delp, PhD, Principal Investigator — Florida State University, College of Medicine; Emily Pritchard, PhD, Principal Investigator — Florida State University, College of Medicine
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No